CLINICAL TRIAL: NCT07380789
Title: Management of Acute Pain After Thoracic Combat Trauma: A Multicenter Study in Ukraine
Brief Title: Comprehensive Multicenter Study on the Management of Acute Pain Following Thoracic Combat-Related Trauma in Ukraine
Acronym: CMS-APT-UA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lviv National Medical University (Other)
Collaborators: Vinnitsa National Medical University (Other)
Responsible Party: Principal Investigator, Maksym Barsa, Medical director, Yuri Semenyuk Rivne Regional Clinical Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPMS-VRL
Record Dates: First submitted 2026-01-17; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pain Management; Thoracic Trauma; Pulmonary Function; Quality of Life; Functional Outcome; Depression in Adults; Neuropathic Pain; Hypoesthesia
Keywords: Acute Pain Management; Thoracic Trauma; Cryoablation; Radiofrequency Ablation; Combat-Related Injury
MeSH Terms: conditions — Agnosia; Neuralgia; Hypesthesia | interventions — Cryosurgery; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryoablation (Active Comparator): Participants assigned to this arm will receive intercostal nerve cryoablation as part of acute pain management following thoracic combat-related trauma. Cryoablation will be performed using a percutaneous, image-guided technique targeting intercostal nerves corresponding to the distribution of thoracic injury. Local cooling will be applied to produce a temporary and reversible interruption of nerve conduction with the aim of reducing pain transmission. The number of intercostal levels treated will be determined based on clinical assessment and injury pattern. Cryoablation will be administered in addition to standard trauma and supportive care according to institutional protocols.
  Interventions: Procedure: Cryoablation
- Radiofrequency Ablation (Active Comparator): Participants assigned to this arm will receive intercostal nerve radiofrequency ablation as part of acute pain management following thoracic combat-related trauma. Radiofrequency ablation will be performed using a percutaneous, image-guided technique targeting intercostal nerves associated with the site of thoracic injury. Controlled radiofrequency energy will be applied to modulate nerve function and reduce pain transmission. The number of intercostal levels treated will be determined based on clinical assessment and injury pattern. Radiofrequency ablation will be administered in addition to standard trauma and supportive care according to institutional protocols.
  Interventions: Procedure: Radiofrequency ablation alone

INTERVENTIONS:
Procedure: Cryoablation — Cryoablation and radiofrequency ablation are minimally invasive interventional pain management techniques used in this study to target intercostal nerves involved in pain transmission following thoracic combat-related trauma. Cryoablation achieves analgesia through the localized application of extreme cold, producing a temporary and reversible interruption of nerve conduction while preserving nerve structure. In contrast, radiofrequency ablation uses controlled radiofrequency-generated thermal energy to modulate nerve function and reduce pain transmission. Both interventions are performed percutaneously under image guidance to ensure accurate targeting of the affected intercostal nerves, with the number of treated levels determined by injury pattern and clinical assessment. Each intervention is administered in addition to standard trauma and supportive care, with the aim of reducing acute pain intensity, limiting opioid requirements, and improving functional outcomes such as respirator
  Arms: Cryoablation
Procedure: Radiofrequency ablation alone — Radiofrequency ablation is a minimally invasive interventional technique that uses controlled radiofrequency-generated thermal energy to modulate peripheral nerve function and reduce pain transmission. In this study, radiofrequency ablation is applied to intercostal nerves associated with thoracic combat-related trauma using a percutaneous, image-guided approach. Thermal energy is delivered in a controlled manner to achieve nerve modulation while limiting damage to surrounding tissues. This intervention is intended to provide effective acute pain relief, reduce opioid requirements, and improve functional outcomes such as respiratory mechanics in patients with thoracic injuries.
  Arms: Radiofrequency Ablation

SUMMARY:
This study is a multicenter clinical trial conducted in Vinnytsia, Rivne, and Lviv, Ukraine, focusing on the management of acute pain following thoracic injuries sustained during combat. The main purpose of the study is to evaluate and compare the effectiveness and safety of two minimally invasive procedures, cryoablation and radiofrequency ablation, in controlling severe chest pain and improving patients' recovery. Cryoablation involves applying extreme cold to specific intercostal nerves to reduce pain signals, while radiofrequency ablation uses controlled heat to achieve a similar effect. Both procedures target the nerves responsible for transmitting pain from the injured areas and are performed by experienced clinicians under careful monitoring to minimize risks. Adult patients who have experienced thoracic combat trauma and are experiencing moderate to severe pain may be eligible to participate in the study if they are able to provide informed consent and comply with the study procedures. Participants will be randomly assigned to receive either cryoablation or radiofrequency ablation. Pain intensity will be assessed before the procedure, and then again at four, twenty-four, and seventy-two hours afterward using a standardized verbal numeric rating scale. In addition to measuring changes in pain, the study will monitor opioid medication use to determine whether either procedure reduces the need for pain-relieving drugs. Mechanical pain sensitivity will be evaluated using Von Frey testing, and pulmonary function will be assessed using incentive spirometry to determine whether pain reduction improves the ability to breathe deeply and cough effectively. The impact of pain on daily activities, quality of life, and emotional well-being will also be measured using validated tools such as the LANS scale, the McGill Pain Questionnaire, and the PHQ-9 depression screening questionnaire. The study aims to provide important information on the relative benefits and risks of cryoablation and radiofrequency ablation for the treatment of acute thoracic pain, including changes in pain intensity, opioid consumption, respiratory function, and overall comfort. Potential risks associated with the procedures include temporary soreness, bruising, or rare complications, but all interventions are performed under strict safety protocols. Participation in this study may allow patients to experience better pain control, potentially reduced reliance on opioid medications, and faster recovery, while contributing valuable data that could improve pain management strategies for other patients in similar circumstances. Data collected during the study will be analyzed to compare the effectiveness of the two procedures and to identify factors that may influence outcomes, such as age, body mass index, the number of intercostal levels treated, and baseline pain scores. The study provides a structured, evidence-based approach to understanding acute pain management after thoracic combat injuries and aims to support clinicians in making informed decisions to improve patient care. For patients, families, and healthcare providers, this research offers an opportunity to participate in a carefully monitored clinical trial designed to enhance recovery and reduce suffering after serious chest trauma while advancing medical knowledge in the field of pain management.

DETAILED DESCRIPTION:
This study is a prospective, multicenter clinical investigation designed to compare cryoablation and radiofrequency ablation as interventional techniques for the management of acute pain following thoracic combat-related trauma in adult patients treated in Ukraine. Thoracic injuries sustained during combat are commonly associated with severe acute pain, which can negatively affect respiratory mechanics, impair coughing and mobilization, increase opioid requirements, and contribute to pulmonary complications and prolonged recovery. Effective and timely pain control is therefore a critical component of trauma care in this patient population.

Cryoablation and radiofrequency ablation are minimally invasive procedures that target peripheral nerves involved in pain transmission, most commonly intercostal nerves in the setting of thoracic trauma. Cryoablation induces a temporary and reversible disruption of nerve conduction through localized application of extreme cold, while radiofrequency ablation produces thermal modulation of nerve function using controlled radiofrequency energy. Both techniques aim to provide targeted analgesia while reducing reliance on systemic analgesics, particularly opioids. Although both approaches are used in clinical practice, comparative evidence regarding their effectiveness, functional impact, and opioid-sparing potential in patients with acute thoracic combat trauma remains limited.

The study will be conducted at multiple tertiary care centers in Vinnytsia, Rivne, and Lviv. Adult patients presenting with thoracic combat-related trauma and clinically significant acute pain will be screened for eligibility and enrolled after providing informed consent. Participants will be randomly assigned to receive either cryoablation or radiofrequency ablation as part of their acute pain management, in addition to standard trauma care according to institutional protocols. The selection of intercostal levels for treatment will be based on injury distribution and clinical assessment, following a standardized procedural approach to ensure consistency across centers.

Pain intensity will be assessed using the Verbal Numeric Rating Scale at baseline prior to intervention and at predefined time points after the procedure to evaluate early and short-term analgesic effects. Opioid consumption will be recorded before intervention and during follow-up and standardized to allow comparison between treatment groups. Because thoracic pain directly affects respiratory function, pulmonary performance will be evaluated using incentive spirometry before and after the intervention to assess changes in airflow and the ability to perform deep breathing and coughing maneuvers.

Mechanical pain sensitivity will be assessed using Von Frey testing to evaluate changes in nociceptive thresholds following treatment. Pain provoked by coughing, a clinically relevant indicator of functional pain control in thoracic trauma, will be measured using a visual analog scale. In addition, patient-reported outcome measures will be collected using validated instruments, including the LANS scale for neuropathic pain features, the McGill Pain Questionnaire for qualitative pain assessment, and the PHQ-9 to screen for depressive symptoms that may influence pain perception and recovery.

Demographic and clinical variables, including age, body mass index, baseline pain severity, and the number of intercostal levels treated, will be collected to support exploratory and adjusted analyses. Data will be entered into a standardized electronic case report form to ensure data quality and consistency across sites. Statistical analyses will include assessment of within-group changes over time and between-group comparisons of pain reduction, opioid use, respiratory function, and patient-reported outcomes. Multivariable analyses may be performed to identify factors associated with treatment response and clinically meaningful pain reduction.

Safety will be monitored throughout the study period. All procedures will be performed by clinicians experienced in interventional pain management techniques, following established institutional and procedural safety standards. Adverse events related to the interventions will be documented and reviewed. Given the acute nature of the intervention and follow-up period, safety assessments will focus on immediate and early procedural complications.

This study aims to generate clinically relevant evidence regarding the comparative effectiveness and safety of cryoablation and radiofrequency ablation for acute pain management following thoracic combat-related trauma. The results are expected to inform clinical decision-making, support optimization of pain management strategies, reduce opioid exposure, and improve functional recovery in this high-risk patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Thoracic trauma from combat-related injuries
* VNRS ≥4 for acute thoracic pain
* Ability to provide informed consent

Exclusion Criteria:

* Severe coagulopathy
* Infection at intervention site
* Allergy to local anesthetics
* Inability to perform spirometry

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4, 24, and 72 hours post-procedure.
  Pain intensity was assessed using the Verbal Numeric Rating Scale (VNRS), a validated 11-point scale ranging from 0 to 10, where 0 indicates "no pain" and 10 indicates "worst imaginable pain." Higher scores represent greater pain intensity (worse outcome). Reduction in pain intensity was evaluated by comparing VNRS scores over time.

SECONDARY OUTCOMES:
Mechanical pain threshold | Before and 72 hours after
  Assess mechanical pain threshold changes using Von Frey test
Opioid consumption | before and 72 hours after ablation
  Compare opioid consumption
Forced Vital Capacity (FVC) | Before and 24 hours after
  Forced Vital Capacity (FVC)
  Pulmonary function was assessed using incentive spirometry by measuring Forced Vital Capacity (FVC), expressed in liters (L). FVC was recorded pre-ablation and post-ablation. Higher values indicate better pulmonary function.
Pain during coughing | Before and 24 hours after
  Pain during coughing was assessed using the Visual Analog Scale (VAS), a continuous scale ranging from 0 to 10, where 0 represents "no pain" and 10 represents "worst imaginable pain." Higher scores indicate greater pain intensity (worse outcome).
Evaluate quality of life and functional outcomes with Leeds Assessment of Neuropathic Symptoms and Signs LANS | 6 month after
  Quality of life and functional outcomes were evaluated using the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) pain scale. LANSS is a validated instrument designed to identify and quantify neuropathic pain and its functional impact. The scale consists of symptom-based questions and sensory examination items, with a total score ranging from 0 to 24. A score of 0 indicates no neuropathic pain features, while a score of 24 indicates the maximum severity of neuropathic pain features. Higher LANSS scores reflect greater neuropathic pain burden, increased functional impairment, and poorer quality of life, representing a worse outcome. Changes in LANSS scores were assessed over the study period to evaluate treatment-related effects.
Quality of life and functional outcomes were evaluated using the McGill Pain Questionnaire (MPQ), | 6 mounth
  Quality of life and functional outcomes were evaluated using the McGill Pain Questionnaire (MPQ), a validated multidimensional instrument assessing the sensory, affective, and evaluative components of pain and their impact on daily functioning. The total Pain Rating Index (PRI) derived from the MPQ ranges from 0 to 78, where 0 indicates no pain-related impact and 78 indicates the maximum pain-related impact. Higher scores represent greater pain intensity and functional impairment, corresponding to poorer quality of life and a worse outcome. Changes in MPQ scores were assessed over the study period to evaluate treatment-related effects.
Quality of life and functional outcomes were evaluated using the Patient Health Questionnaire-9 (PHQ-9) | 6 mounth
  Quality of life and functional outcomes were evaluated using the Patient Health Questionnaire-9 (PHQ-9), a validated self-reported instrument used to assess the severity of depressive symptoms and their impact on daily functioning and overall quality of life. The PHQ-9 total score ranges from 0 to 27, where 0 indicates no depressive symptoms and 27 indicates severe depressive symptoms. Higher scores represent greater symptom severity, increased functional impairment, and poorer quality of life, corresponding to a worse outcome. Changes in PHQ-9 scores were assessed over the study period to evaluate treatment-related effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Communal enterprise "Yuri Semenyuk Rivne Regional Clinical Hospital" of Rivne Regional Council, Rivne, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dmytriiev D, Liu W, Barsa M, Khomenko A, Strokan A, Pasquina PF, Cohen SP. Perineuromal hydrodissection for acute postamputation pain? An observational study in a time of war. Reg Anesth Pain Med. 2025 Feb 26:rapm-2024-106307. doi: 10.1136/rapm-2024-106307. Online ahead of print. PMID 39971386
- See also: Related Info — https://uaratb.org/en